CLINICAL TRIAL: NCT04602611
Title: A Randomized, Controlled Prospective Trial Evaluating The Impact Of A Nurse Navigation Program on Patients With Gastrointestinal Cancers Undergoing Oncological Treatment
Brief Title: Impact Of Nurse Navigation Program on Outcomes in Patients With GI Cancers
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00081349.; 00046658; LCI-GI-NOS-NAV-001 (Other: Atrium)
Record Dates: First submitted 2020-10-14; First posted 2020-10-26 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care
- Oncology Nurse Navigation (Experimental): Standard of Care + Oncology Nurse Navigation
  Interventions: Other: Oncology Nurse Navigation

INTERVENTIONS:
Other: Oncology Nurse Navigation — Providing the subject with the service of navigation (ONN) performed under LCI Patient Navigation Program (LPNP), led by a registered oncology nurse.
  Arms: Oncology Nurse Navigation

SUMMARY:
The purpose of this study is to learn about the impact of the Oncology Nurse Navigation program on the frequency of Emergency Department, urgent care visits and inpatient hospital admissions; and overall survival rate at 6 months. The investigators aim to understand if prompt and effective coordination of care provided by Oncology Nurse Navigation (ONN) service will reduce the number of avoidable, unplanned ED visits and hospitalizations, as well as adding measurable value to cancer care, and improve patient overall survival.

DETAILED DESCRIPTION:
A randomized controlled prospective trial evaluating the effectiveness of a nurse navigation program for gastrointestinal cancer patients undergoing oncological treatment. Upon accrual, patients will be randomized 1:1 to receive standard of care plus ONN service (n = 107) or standard of care only (without ONN service; n = 107). Patients in both arms will be assessed for acute care utilization and overall survival (OS) rate at 6 months. Anticipated accrual period will be 30 months.

ELIGIBILITY:
Inclusion Criteria

1. Informed consent and HIPAA authorization for the release of personal health information
2. Aged ≥ 18 years at the time of consent
3. Subject is planning to receive their cancer care at LCI at the time of consent
4. Treatment naïve OR adjuvant greater than 6 months ago, histologically or cytologically confirmed one of the following diagnoses (metastatic/recurrent status can be radiologically confirmed):

   1. Metastatic/recurrent or locally advanced, unresectable or borderline resectable (as defined per NCCN, Alliance or other acceptable guidelines criteria) pancreatic cancer
   2. Metastatic/recurrent or locally advanced, unresectable esophageal, gastroesophageal junction (GEJ) or gastric cancer patients or those who are not eligible for surgery
   3. Metastatic/recurrent or locally advanced, unresectable hepatocellular carcinoma (HCC)

      * radiographic confirmation of the HCC diagnoses is acceptable
      * prior locoregional treatment for subjects with HCC is allowed, but no prior systemic therapy is allowed
   4. Metastatic/recurrent or advanced, unresectable biliary cancers (e.g. gall bladder cancer, cholangiocarcinoma)

      • prior locoregional treatment for subjects with biliary cancers is allowed, but no prior systemic therapy is allowed
   5. Metastatic colorectal or small bowel cancer patients who had disease progression on or are intolerant to fluorouracil/capecitabine, oxaliplatin, and irinotecan-based therapy (e.g. FOLFOX, FOLFIRI or FOLFOXIRI)

      * Subjects can be enrolled within, but no later than 30 days after initiation of their systemic therapy, however every effort will be made to enroll subjects prior to the initiation of systemic therapy. Subjects who has completed or undergoing a current palliative radiotherapy are allowed
5. Ability to read and understand the English or Spanish language
6. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study. However, refusal to complete a patient satisfaction questionnaire IL109 should not refrain a subject from being enrolled.
7. Life expectancy is > 3 months

Exclusion Criteria

1. Subjects have previously received or are currently receiving LCI Patient Navigation Program services
2. Subjects with colorectal cancer enrolled in the Empower Program
3. Subjects with low grade neuroendocrine tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Salem, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Oncology Nurse Navigation
Started (Randomized/Enrolled) | 115 | 113
Completed (Off study) | 115 | 113
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Oncology Nurse Navigation | Total
Number analyzed (Participants) | 115 | 113 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 52 | 51 | 103
  >=65 years | 63 | 61 | 124
Age, Continuous [Median (Full Range); unit: years] | 66 [29 to 91] | 65 [18 to 88] | 66 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 52 | 86
  Male | 81 | 61 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 106 | 111 | 217
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 30 | 56
  White | 85 | 80 | 165
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 115 | 113 | 228
Diagnosis [Count of Participants; unit: Participants]
  Colorectal cancer (progression on or intolerant to fluorouracil, oxaliplatin and irinotecan therapy) | 6 | 4 | 10
  Locally advanced unresectable pancreatic cancer | 16 | 16 | 32
  Metastatic or unresectable biliary cancer | 16 | 16 | 32
  Metastatic or unresectable gastroesophageal cancer | 21 | 20 | 41
  Metastatic or unresectable hepatocellular carcinoma | 15 | 16 | 31
  Metastatic pancreatic | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Annualized Count of Acute Care Visits
Description: The annualized count of acute care visits, where acute care visits included all unplanned inpatient admissions, emergency room encounters, and/or urgent care visits, was calculated for each subject as the total number of acute care visits normalized to an annual basis.
Time Frame: From the date of randomization until subject discontinued the intervention, assessed up to 34 months
Population: Enrolled participants who both (a) received at least one dose of standard of care systemic anti-cancer therapy on or after the enrollment date and (b) died within six months of enrollment or otherwise were on study for at least 6 months.
Measure: Median (Inter-Quartile Range); unit: unplanned acute care visits in one year
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 87 | 95
unplanned acute care visits in one year | 3 [0 to 9.6] | 3.8 [1.3 to 7.7]
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; The study was designed with co-primary objectives evaluating acute care utilization (ACU) and 6-month OS rate. Power/sample size were calculated based on the OS objective. The overall type I error rate was alpha=0.05; the co-primary objectives were powered at the 2-sided alpha=0.025 significance level. Three hundred evaluable subjects would have provided >=93% power to detect a 20% reduction in ACU (assuming there were 6 ACUs per year in SOC arm). The study did not achieve targeted enrollment; Test type: Superiority; p = 0.80, Regression, Negative binomial — The a priori threshold for statistical significance was 0.025; Model was estimated without adjustments (sole covariate was treatment; coefficient was the estimated treatment effect) using 180 degrees of freedom; Coefficient of negative binomial model = 0.0547, 95% CI 2-sided [-0.3680 to 0.4773] — The estimated coefficient was associated with Oncology Nurse Navigation with reference to Standard of Care

2. Primary Outcome: Proportion of Participants Surviving at 6 Months
Description: The proportion of participants surviving at 6 months was calculated for each treatment arm. Six-month overall survival was determined for each subject as a binary variable indicating whether or not the subject was alive at 6 months after study enrollment. Failure occurred if the subject died from any cause within 6 months of study enrollment. The proportions were compared between the arms.
Time Frame: From the date of randomization to death or 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 87 | 95
Participants | 52 | 58
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.88, Fisher Exact — The a priori threshold for statistical significance was 0.025; No adjustments were made in this analysis; The proportions of evaluable subjects surviving at 6 months were analyzed in a 2x2 contingency table using Fisher's Exact test. In the SOC arm, 52/87(60%) evaluable subjects were alive at 6 months and 35/87 (40%) were not. In the ONN + SOC arm, 58/95 (61%) evaluable subjects were alive at 6 months and 37/95 (39%) were not. The p-value estimated using Fisher's Exact test on this 2x2 contingency table was p=0.88

3. Secondary Outcome: Proportion of Participants Surviving at 12 Months
Description: The proportion of participants surviving at 12 months was calculated for each treatment arm. Six-month overall survival was determined for each subject as a binary variable indicating whether or not the subject was alive at 12 months after study enrollment. Failure occurred if the subject died from any cause within 12 months of study enrollment. The proportions were compared between the arms.
Time Frame: From the date of randomization up until 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 87 | 95
Participants | 23 | 28
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p = 0.74, Fisher Exact — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; No adjustments were made in this analysis; The proportions of evaluable subjects surviving at 12 months were analyzed in a 2x2 contingency table using Fisher's Exact test. In the SOC arm, 23/87(26%) evaluable subjects were alive at 12 months and 64/87(74%) were not. In the ONN + SOC arm, 28/95 (29%) evaluable subjects were alive at 6 months and 67/95 (71%) were not. The p-value estimated using Fisher's Exact test on this 2x2 contingency table was p=0.74

4. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay was calculated for each subject as the total number of unplanned inpatient days while on intervention.
Time Frame: From the date of randomization until subject discontinued the intervention, assessed up to 34 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 87 | 95
Days | 1 [0 to 10] | 4 [0 to 92]
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p = 0.57, Regression, Negative binomial — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; [statistical method as in outcome 1, analysis 1]; Coefficient of negative binomial model = 0.1574, 95% CI 2-sided [-0.3905 to 0.7054] — The estimated coefficient was associated with Oncology Nurse Navigation with reference to Standard of Care

5. Secondary Outcome: Time From Hospice Referral to Death for Participants Referred to Hospice
Description: Time from hospice referral to death was a time-to-event endpoint defined as the time from hospice referral to the date of death from any cause. Subjects who were alive or lost to follow-up at the time of the analysis were censored at the last known date they were alive. This endpoint was only calculated for subjects referred to hospice.
Time Frame: From the date of hospice referral to death or last follow-up, assessed over 7 months.
Population: Enrolled participants who both (a) received at least one dose of standard of care systemic anti-cancer therapy on or after the enrollment date, (b) died within six months of enrollment or otherwise were on study for at least 6 months, and (c) were referred to hospice (82/228 participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 39 | 43
months | 0.427 [0.263 to 0.755] | 0.526 [0.296 to 1.084]
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p = 0.45, Log Rank — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; Unadjusted log-rank test; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.570 to 1.309] — The estimated hazard ratio was associated with Oncology Nurse Navigation with reference to Standard of Care; the model was estimated without adjustments (the sole covariate was treatment)

6. Secondary Outcome: Total Number of 30-day Readmissions
Description: The number of readmissions within 30 days of in-patient admission discharges was calculated for each participant. This outcome was derived for each subject with at least one in-patient admission.
Time Frame: From the date of randomization until subject discontinued the intervention, assessed up to 34 months
Population: Enrolled participants who both (a) received at least one dose of standard of care systemic anti-cancer therapy on or after the enrollment date, (b) died within six months of enrollment or otherwise were on study for at least 6 months, and (c) had at least one in-patient admission (115/228 participants).
Measure: Median (Inter-Quartile Range); unit: number of 30-day readmissions
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 51 | 64
number of 30-day readmissions | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p = 0.21, Regression, Negative binomial — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; [statistical method as in outcome 1, analysis 1]; Coefficient of negative binomial model = -0.4194, 95% CI 2-sided [-1.0763 to 0.2374] — The estimated coefficient was associated with Oncology Nurse Navigation with reference to Standard of Care

7. Secondary Outcome: Proportion of Participants Referred to Supportive Care Services
Description: Referral to Supportive Care Services was derived for each participant as a binary variable indicating if there was at least one documented referral to Palliative Care, Nutrition Services, and/or Social Work Services.
Time Frame: From the date of randomization until subject discontinued the intervention, assessed up to 34 months
Population: Enrolled participants who both (a) receive at least one dose of standard of care systemic anti-cancer therapy on or after the enrollment date and (b) die within six months of enrollment or otherwise are on study for at least 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 87 | 95
Participants | 22 | 50
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p < 0.01, Regression, Logistic — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; Model was estimated without adjustments (the sole covariate was treatment); Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.75 to 6.15] — The estimated odds ratio was associated with Oncology Nurse Navigation with reference to Standard of Care

8. Secondary Outcome: Proportions of Missed Visits of All Scheduled Visits From 0% to 100%.
Description: This proportion was calculated for each participant as the percentage of missed visits of all scheduled within Atrium Health, regardless of visit type.
Time Frame: From the date of randomization until subject discontinued the intervention, assessed up to 34 months
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of missed scheduled visits
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 87 | 95
percentage of missed scheduled visits | 3.1 [0.0 to 47.6] | 2.2 [0.0 to 60.0]
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p = 0.11, Regression, Linear — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; Model was estimated without adjustments (sole covariate was treatment; slope was the estimated treatment effect) using 180 degrees of freedom; Slope = -2.6939, 95% CI 2-sided [-5.9538 to 0.5659] — The estimated slope was associated with Oncology Nurse Navigation with reference to Standard of Care

9. Secondary Outcome: Average Score of Subject Satisfaction as Assessed by an Adaptation of the EORTC PATSAT C33
Description: Subject satisfaction was assessed by a modified European Organization for Research and Treatment of Cancer Patient Satisfaction with cancer care questionnaire #33 (EORTC PATSAT C33) 10-14 weeks after randomization. Subjects completed the questionnaire assessing thirty-four elements of their experience with regards to hospital environment, hospital personnel, and treatment. Each question was assessed on a Likert-type scale ranging Poor to Excellent (mapped numerically to 1-5), where the higher scores indicated a better experience. The average score was calculated for each subject as the sum of the non-missing standardized scores divided by the number of measures contributing to the sum. The average score could range from 1 (the minimum) to 5 (the maximum).
Time Frame: From the date of randomization up until 14 weeks
Population: Enrolled participants who both (a) received at least one dose of standard of care systemic anti-cancer therapy on or after the enrollment date, (b) died within six months of enrollment or otherwise were on study for at least 6 months, and (c) completed the subject satisfaction survey 10-14 weeks after randomization (86/228 participants).
Measure: Mean (Standard Deviation); unit: score on a scale (out of 5)
Arm/Group | Standard of Care | Oncology Nurse Navigation
Number analyzed (Participants) | 35 | 51
score on a scale (out of 5) | 4.4 (0.6) | 4.6 (0.5)
Statistical Analysis 1: Comparison: Standard of Care vs Oncology Nurse Navigation; Test type: Superiority; p = 0.09, Regression, Linear — This p-value was not adjusted for multiple comparisons; the a priori threshold for statistical significance was p=0.05; This univariate model was not adjusted for other covariates; this model was estimated using 84 degrees of freedom; Slope = 0.1197, 95% CI 2-sided [-0.0315 to 0.4378] — The estimated slope was associated with Oncology Nurse Navigation with reference to Standard of Care

ADVERSE EVENTS:
Time Frame: From the date of randomization until subject discontinued study involvement, assessed up to 34 months
Description: The number of participants who died while on study is summarized. Other adverse events were not collected for study purposes as the intervention was unlikely to present harm to enrolled participants above standard of care.
  The number of participants at risk for Serious Adverse Events is zero because adverse events were not monitored/assessed.
  The number of participants at risk for Other (Not Including Serious) Adverse Events is zero because adverse events were not monitored/assessed.
Arm/Group | Standard of Care | Oncology Nurse Navigation
All-Cause Mortality (participants affected / at risk) | 72/115 | 77/113
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04602611/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04602611/ICF_000.pdf